CLINICAL TRIAL: NCT04024826
Title: Acute Effects of Resistance Training on Substrate Metabolism During Different Phases of Menstrual Cycle
Brief Title: Effects of Resistance Training on Substrate Metabolism During the Menstrual Cycle
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid/19
Sponsor: Southern Illinois University Edwardsville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 111A
Record Dates: First submitted 2019-03-21; First posted 2019-07-18 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2019-07

CONDITIONS: Menstrual Cycle; Substrate Metabolism
Keywords: resistance training; carbohydrate metabolism; fat oxidation

STUDY DESIGN:
Intervention Model Description: The participants will be randomized into either one of the 4 four phases- namely Early Follicular Phase(EFP-Days1 to 7), Late Follicular Phase(LFP-Days 8 to 14), Early Luteal Phase(ELP-Days 15 to 21) or Late Luteal Phase(LLP-Days 22 to 28) of the menstrual phase. Once the participant is assigned to one of the phases. Each participant will undergo 4 intervention days. the first intervention day will take place during the mid-point of the said phase i.e. EFP- Day 4. After one intervention is complete there will be a washout period and the intervention will take place on the 7th day after the first intervention i.e if the first intervention is LFP done on day 11 of the menstrual cycle the next intervention will take place on day 18 of menstrual cycle which will account for ELP. In this manner, the Participant will be tested in all 4 phases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Follicular Phase (EFP) (Experimental): This group is comprised of participants at the Early Follicular Phase (EFP) of the menstrual cycle.
  Interventions: Behavioral: EFP
- Late Follicular Phase (Experimental): This group is comprised of participants at the Late Follicular Phase (LFP) of the menstrual cycle.
  Interventions: Behavioral: LFP
- Early Luteal Phase (Experimental): This group is comprised of participants at the Early Luteal Phase (ELP) of the menstrual cycle.
  Interventions: Behavioral: ELP
- Late Luteal Phase (Experimental): This group is comprised of participants at the Late Luteal Phase(LLP) of the menstrual cycle.
  Interventions: Behavioral: LLP

INTERVENTIONS:
Behavioral: EFP — This group will perform the Resistance training intervention on day 4 of the menstrual cycle, which corresponds to the mid of early follicular phase.
  Arms: Early Follicular Phase (EFP)
Behavioral: LFP — This group will perform the Resistance training intervention on day 11 of the menstrual cycle, which corresponds to the mid of late follicular phase.
  Arms: Late Follicular Phase
Behavioral: ELP — This group will perform the Resistance training intervention on the day 18 of the menstrual cycle, which corresponds to the mid of early luteal phase
  Arms: Early Luteal Phase
Behavioral: LLP — This group will perform the Resistance training intervention on day 21 of the menstrual cycle, which corresponds to the mid of late luteal phase
  Arms: Late Luteal Phase

SUMMARY:
This research project's objective is to investigate substrate metabolism behavior in response to the RT during different phases of the menstrual cycle.

DETAILED DESCRIPTION:
Based on the literature the investigators hypothesize an increase in fat oxidation in early follicular phase(EFP) and late follicular phase (LFP) when compared to early luteal phase (ELP) and late luteal phase (LLP). Given the lack of research in exercise and menstrual cycle - especially in resistance training - results are uncertain unless the investigators base their hypotheses only on the general physiological effects of sex hormones (without exercise). In this case, the investigators expect to see a reduced carbohydrate utilization and an increased utilization of fats in EFP and LFP. In addition, the intervention is focused on muscular endurance and, therefore, it is expected to see a higher reliance on aerobic pathways. It is expected that the effects of the intervention will be added to the effects of estrogens, with increasing fat oxidation when estrogen levels are higher. Lastly, a comparison of fat oxidation levels obtained on each sub-phase would reveal if there are differences in the magnitude of the effect of distinct concentrations of estrogen and progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Females with BMI-18.5-34.99 and between 18-45 years, with normal menstrual cycle defined as 28-30 days cycles +-3 days.
* Including higher BMI participants might alter the results as increased body fat has been linked to changes in different hormonal levels (not only sex hormones) and that might influence substrate utilization.
* Sedentary .or physically active for 2 days a week or less.

Exclusion Criteria:

* • Musculoskeletal injuries,

  * cardio-respiratory conditions,
  * metabolic conditions,
  * irregular menstrual cycle,
  * menstrual dysfunction or unusual sex hormone levels,
  * on contraceptives,
  * on medication that alter hormonal or cardio-respiratory responses,
  * pre-menopausal symptoms,
  * on moderate to high-intensity exercise regime more than 2d/week.
  * All these exclusion criteria are chosen because any one of the listed criteria above can alter the responses and/or affect the safety of the subject during their participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females with a normal menstrual cycle defined as 28-30 days and a duration of 3-7 days with BMI-18.5-34.99 and between 18-45 years.
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Changes in Substrate oxidation | During each exercise session: 1 assessment point on each menstrual cycle phase
  changes in substrate oxidation will be measured using cosmed K5 during the intervention phase
Changes in Estrogen levels. | At baseline: 1 assessment point on each menstrual cycle phase
  Blood would be drawn from the participants for assessment of hormone estrogen
Changes in Progesterone levels. | At baseline: 1 assessment point on each menstrual cycle phase
  Blood would be drawn from the participants for assessment of hormone Progesterone.

SECONDARY OUTCOMES:
Muscular strength | At baseline: 1 assessment point
  Muscular strength will be assessed by one-repetition maximum test on leg press and bench press
Cardiorespiratory Function | At baseline: 1 assessment point
  maximal oxygen consumption will measured on a treadmill with a metabolic cart
Relative Body Fat (%) | At baseline: 1 assessment point
  Body composition i.e Fat mass, Lean body mass and Body fat percentage will be measured using dual-energy xray absorptiometry
Lean Body Mass (kg) | At baseline: 1 assessment point
  Body composition i.e Fat mass, Lean body mass and Body fat percentage will be measured using dual-energy xray absorptiometry
Fat Mass (kg) | At baseline: 1 assessment point
  Body composition i.e Fat mass, Lean body mass and Body fat percentage will be measured using dual-energy xray absorptiometry
Diet | At baseline: 1 assessment point on each menstrual cycle phase
  Diet will be measured using ASA-24h recall

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Southern Illinois University Edwardsville
Locations (1):
- Southern Illinois University Edwardsville, Edwardsville, Illinois, United States